CLINICAL TRIAL: NCT03841318
Title: Involvement of Immune Cells Derived From the Intestine in Sjogren's Syndrome
Acronym: SINGOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2018/53
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Sjogren's Syndrome
Keywords: lymphoid cells; gut-derived lymphocytes
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sjogren's Syndrome (Experimental)
  Interventions: Biological: blood sample; Biological: biopsy of the labial salivary gland

INTERVENTIONS:
Biological: blood sample — 36 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Biological: biopsy of the labial salivary gland — Part of the biopsy of the labial salivary gland

SUMMARY:
The study aims at defining the role of immune cells derived from the intestine in the pathogenesis of Sjogren's disease. This research might open new therapeutic approaches for the treatment of autoimmune diseases.

DETAILED DESCRIPTION:
Autoimmune diseases are characterized by a loss of tolerance of the immune system for self-antigens. One of the feature of autoimmune diseases is the infiltration of lymphoid cells in the tissues damaged by the disease (i.e. kidney in systemic lupus erythematous or brain in multiple sclerosis). However, the origins and properties of the immune cells infiltrating these target tissues are largely unknown.

Studies in mouse models have shown that the composition of the gut microbiota can modify the susceptibility to autoimmune diseases. These studies demonstrated that the microbiota composition can alter the pathogenic properties of T cells in the gut but also in the target tissues. For instance, in the experimental autoimmune encephalomyelitis model, the composition of the gut microbiota has been shown to modulate the susceptibility to the disease and the properties of the pathogenic CD4 T cells in the gut but also in the central nervous system. In human an alteration in the composition of the gut microbiota is observed in numerous autoimmune diseases, including Sjogren's syndrome, suggesting that perturbation of the gut microbiota might be linked to the pathogenicity of immune cells in the target organs. However, the mechanisms by which the microbiota impacts the pathogenicity of immune cells in the target organs is unknown. It is proposed that gut immune cells directly exposed to the microbiota compounds could migrate to the target organs and participate to the buildup of tissue damages. This hypothesis is supported by studies in mouse models showing the migration of gut CD4 T cells in the inflamed kidney (glomerulonephritis model) or in the systemic lymphoid organs (rheumatoid arthritis model). The preliminary data support this hypothesis as the investigators have shown that gut-derived CD4 T cells display pathogenic properties in human autoimmune diseases. To determine whether and how the gut-derived immune cells are involved in the pathogenesis of autoimmune disease, the investigators propose to study the origin and properties of immune cells infiltrated in target tissues in autoimmune diseases.

Sjogren's syndrome is a systemic autoimmune disease in which exocrine gland in particular lacrimal and salivary glands are affected. One of the hallmark of the disease is the infiltration of lymphoid cells in the exocrine glands of the patients. Indeed, the presence of lymphoid infiltrate in the minor labial salivary gland of the patients is one of the most important diagnostic tool for Sjogren's syndrome. The investigation of lymphoid infiltrates requires to perform a biopsy of the labial salivary gland. The investigators propose here to take advantage of this minimally invasive procedure to study the properties of the lymphoid cells present in the minor salivary glands of Sjogren's patients.

The study will recruit 200 patients followed in Bordeaux University Hospital in which a salivary gland biopsy is performed for a clinical suspicion of Sjogren's syndrome. Blood and a biopsy of the minor salivary gland of the lip will be collected during a scheduled visit to study the properties of infiltrated immune cells. Clinical and biological disease activity, treatment and outcomes will be studied in correlation with the properties of infiltrated immune cells. No extra visit will be needed and the biopsy of the minor salivary gland of the lip and the blood samples will be collected at the same times as those collected for clinical purposes.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of Sjogren's syndrome based on 2016 American College of Rheumatology (ACR) criteria;
* Age ≥ 18 years
* Being affiliated to health insurance
* Willing to participate

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Quantification of the immune cells infiltrated in the minor salivary glands of Sjogren's patients. | At baseline (Day 0)

SECONDARY OUTCOMES:
Quantification of disease activity scores for Sjogren's patients evalued by EULAR Sjögren Syndrome Disease Activity Index | At baseline (Day 0)
  EULAR Sjögren Syndrome Disease Activity Index (ESSDAI) : between 0 and 123, in which higher values indicate higher severity

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DUFFAU, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Service de médecine interne, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No